CLINICAL TRIAL: NCT03569787
Title: A Retrospective Cohort Study of Hyperprolactinaemia Management in Reproductive Services at University Hospital of Coventry and Warwickshire (UHCW)
Brief Title: Hyperprolactinaemia Management in Reproductive Services at University Hospital of Coventry and Warwickshire
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GF0253
Record Dates: First submitted 2018-04-30; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Hyperprolactinemia; Subfertility; Subclinical hypothyroïdism
MeSH Terms: conditions — Hyperprolactinemia; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hyperprolactinaemia: Patients undergoing subfertility studies with at least one high prolactin reading (>500mU/L).
  Interventions: Diagnostic Test: MRI Pituitary

INTERVENTIONS:
Diagnostic Test: MRI Pituitary — Identification of whether of not patients had had an MRI pituitary following hyperprolactinaemia reading

SUMMARY:
Hyperprolactinaemia and thyroid disorders can significantly reduce fertility by causing ovulatory dysfunction. There is no evidence to suggest treatment of hyperprolactinaemia in the presence of regular ovulatory menstruation will improve fertility. However, anecdotal observation of practice at UHCW NHS Trust suggested that dopamine agonists are often prescribed irrespective of whether symptoms of hyperprolactinaemia are present.

The aim of the study was to establish the prevalence of hyperprolactinaemia and incidence of subclinical hypothyroidism in patients undergoing subfertility investigations at UHCW NHS Trust. Also, to examine management of patients with hyperprolactinaemia and a normal pituitary MRI scan, and explore the trends in treatment; and finally, to explore how this could improve reproductive services.

107 patients were identified as having a high prolactin reading between January 2014 and January 2017. Hospital records were examined for patient demographics, relevant blood and scan results, medical history, any treatment, and treatment outcomes.

The prevalence of hyperprolactinaemia was 23%. 20.6% of patients had suboptimal thyroid function and were started on levothyroxine. Prolactin levels, and presence of relevant symptoms, only had a partial bearing on whether dopamine agonists were used in those with normal pituitary MRI results (or where no scan was performed). The use of dopamine agonists appeared to correlate with assisted conception and a lower incidence of birth complications (inc. miscarriage, prematurity), though the significance of this was limited by the size of the dataset.

Dopamine agonists often appeared to be used in more complex patients, rather than exclusively those with a higher prolactin reading and/or the presence of related symptomatology. Patients frequently underwent a pituitary MRI scan in the absence of symptoms, contrary to evidence. The findings suggest that less patients should be scanned and less treated with dopamine agonists. A health economics evaluation study would be useful to elucidate the potential cost saving this could represent. It may be better to prioritise optimisation of thyroid function, particularly when noting the similarities in the prevalence of suboptimal thyroid function and that of hyperprolactinaemia.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing care through subfertility services at UHCW
* Referred and seen in subfertility services between January 2014 to October 2017
* Identified as having had at least one episode of hyperprolactinaemia within the study period (Jan 2014 to January 2017)

Exclusion Criteria:

* Referred outside of study period
* Hyperprolactinaemia reading outside of study period

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients seen in subfertility services at UHCW between January 2014 to October 2017
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Number of people referred to subfertility services identified as having at least one high serum prolactin result (>500mU/L) as identified by UHCW CRRS (University Hospital of Coventry and Warwickshire Clinical Records Reporting System) records | January 2014 - January 2017
  Not to date of study start to allow period to follow up on conception and birth data
Number of patients who received a course of dopamine agonist (of any length, at any point during access to subfertility services) as identified by UHCW CRRS (University Hospital of Coventry and Warwickshire Clinical Records Reporting System) records | January 2014 - January 2017
  This typically included bromocriptine or cabergoline. Whether or not they were concurrently treated with Levothyroxine was also recorded (either for new subclinical hypothyroidism or coexisting previously diagnosed hypothyroidism).
Number of patients who received a pituitary MRI scan, and the reported result, as identified by UHCW CRRS records | January 2014 - October 2017

SECONDARY OUTCOMES:
Demographics of the mother, including: age at referral, BMI at referral, ethnicity, whether primary or secondary subfertility, previous parities, smoking status, any recorded alcohol consumption as identified by UHCW CRRS records | January 2014 - October 2017
Demographics of father, including: smoking status, any alcohol consumption, semen analysis result, whether the father is receiving treatment for improving semen quality as identified by UHCW CRRS records | January 2014 - October 2017
Relevant blood results for mother (outlined in desciption), as close as possible to referral date to subfertility services as identified by UHCW CRRS records | January 2014 - October 2017
  Including: anti-mullerian hormone (mU/L); oestrodiol; FSH (IU/L); LH (IU/L); testosterone (nmol/L); SHBG; androstenedione; TSH (mU/L); free T4 (pmol/L); TPO antibodies; TSH receptor antibodies; macroprolactin (where negative is more than 50% recovery following PEG test)
Number of patients who experienced symptoms of hyperprolactinaemia, namely any record of: amenorrhoea, oligomenorrhoea, galactorrhoea (inc. whether unilateral or bilateral) and any other relevant symptoms recorded as identified by UHCW CRRS records | January 2014 - October 2017
Number of patients identified as having PCOS, including what elements of the Rotterdam Criteria led to diagnosis as identified by UHCW CRRS records | January 2014 - October 2017
Number of patients with pre-exisitng thyroid disorder, any past medical history, and/or any concomitant medications as identified by UHCW CRRS records | January 2014 - October 2017
Number of patients that managed to conceive, if this was spontaneous (and if not, by what method of assistance), and the outcome of the pregnancy as identified by UHCW CRRS records | January 2014 - October 2017
  Outcome of pregnancy categorised by: birth at term, premature birth, miscarriage, stillbirth or ectopic

CONTACTS AND LOCATIONS:
Locations (1):
- Megan Crowe, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No